CLINICAL TRIAL: NCT01640340
Title: Pilot Study on the Efficacy of an Ondansetron Versus Palonosetron-containing Antiemetic Regimen Prior to Highly Emetogenic Chemotherapy(HEC).
Brief Title: Ondansetron Versus Palonosetron Antiemetic Regimen Prior to Highly Emetogenic Chemotherapy(HEC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Rachel Layman, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-10118; NCI-2012-01009 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-10; First posted 2012-07-13 (Estimated); Results first posted 2013-10-07 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-10

CONDITIONS: Malignant Neoplasm
Keywords: ondansetron; palonosetron; emetogenic chemotherapy; HEC
MeSH Terms: conditions — Neoplasms | interventions — Aprepitant; Palonosetron; Ondansetron; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (palonosetron hydrochloride) (Experimental): Patients receive palonosetron hydrochloride IV 30 minutes prior to chemotherapy on day 1, aprepitant PO (by mouth) 60 minutes prior to chemotherapy on days 1-3, and dexamethasone PO 30 minutes prior to chemotherapy on days 1-4.
  Interventions: Drug: aprepitant; Drug: palonosetron hydrochloride; Drug: dexamethasone
- Arm II (ondansetron) (Experimental): Patients receive ondansetron PO 30 minutes prior to chemotherapy on day 1 and aprepitant and dexamethasone as in Arm I.
  Interventions: Drug: aprepitant; Drug: ondansetron; Drug: dexamethasone

INTERVENTIONS:
Drug: aprepitant — Given by mouth
  Other Names: Emend; L-754030; MK-0869; ONO-7436
Drug: palonosetron hydrochloride — Given IV(intervenous infusion)
  Other Names: Aloxi; RS 25259-197
  Arms: Arm I (palonosetron hydrochloride)
Drug: ondansetron — Given PO
  Other Names: GR 38032F; GR-C507/75; Zofran
  Arms: Arm II (ondansetron)
Drug: dexamethasone — Given PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM

SUMMARY:
Palonosetron is different from ondansetron because it stays in the body longer and may prevent nausea and vomiting for a longer period of time than ondansetron. It is standard practice to use dexamethasone and aprepitant with either ondansetron or palonosetron to prevent nausea and vomiting caused by highly emetogenic chemotherapy. Although these combinations are commonly used, they have never been compared to each other. The purpose of this study is to record the amount of nausea and vomiting, and the amount of "rescue" medication that is used with these two different anti-emetic regimens

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The goal of this study is to evaluate the overall complete response rate (CR, no emesis and no use of rescue medication from 0 to 120 hours after chemotherapy) of two different antiemetic regimens (palonosetron + aprepitant + dexamethasone and ondansetron + aprepitant + dexamethasone) for patients undergoing the first cycle of highly emetogenic chemotherapy (HEC).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive palonosetron hydrochloride intravenously (IV) 30 minutes prior to chemotherapy on day 1, aprepitant orally (PO) 60 minutes prior to chemotherapy on days 1-3, and dexamethasone PO 30 minutes prior to chemotherapy on days 1-4.

ARM II: Patients receive ondansetron PO 30 minutes prior to chemotherapy on day 1 and aprepitant and dexamethasone as in Arm I.

After completion of study treatment, patients are followed up for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed malignancy
* Chemotherapy naive or treated with only low or minimally emetogenic chemotherapy in the past (as defined by the National Comprehensive Cancer Network version [v].2.201 Antiemetic Guidelines)
* Scheduled to receive the first dose of their first cycle of HEC
* Patients receiving multi-day chemotherapy, the HEC portion must be on day 1 and the remaining days of chemotherapy must be minimally emetogenic (i.e. fluorouracil)
* Performance status of Eastern Cooperative Oncology Group (ECOG) grade 0-2
* Able to provide informed consent
* Able to read and write in English or have someone that can that can translate to them and record their diary entries
* Able to take oral medications
* Patients are allowed to participate in a concurrent clinical trial, if the other trial:

  * Does not mandate an antiemetic regimen that interferes with this study
  * Allows antiemetic administration at the physician's discretion
  * Does not prohibit the patient from participating in this study
* Patients must be willing to participate with daily diary entries for 5 days following chemotherapy, and agree to have a 5 minute follow-up call on day 2 or 3 and day 5, 6 or 7

Exclusion Criteria:

* Has stage IV (metastatic) disease
* Known hypersensitivity to ondansetron, palonosetron, aprepitant, or dexamethasone
* Have received or will receive agents that are strong cytochrome P450 3A4 (CYP450 3A4) inducers and/or inhibitors and known to cause clinically relevant drug interactions within one week prior to study treatment and continuing through day 5; any vomiting or retching within 24 hours before administration of chemotherapy
* Grade 2 nausea or greater, according to the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v 4.0) within 24 hours before administration of chemotherapy
* Received an antiemetic within 24 hours before study drug administration, excluding the use of benzodiazepines
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2.5 times upper limit of normal
* Total bilirubin > 1.5 times upper limit of normal

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Layman, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for eligibility during routine clinic visits by a physician, nurse practitioner or pharmacist involved in their care.
Pre-assignment Details: Patients were stratified based upon their chemotherapy regimen (cisplatin versus noncisplatin containing) and then randomized to the ondansetron or palonosetron group.
Groups:
- Arm A (Palonosetron 0.25 mg IV on Day 1): Palonosetron 0.25 mg day 1; aprepitant 125 mg day 1, 80 mg days 2-3; dexamethasone 12 mg day 1, 8 mg day 2-4
- Arm B (Ondansetron 24 mg Oral on Day 1): Ondansetron 24 mg day 1; aprepitant 125 mg day 1, 80 mg day 2-3; dexamethasone 12 mg day 1, 8 mg day 2-4
Period: Overall Study
Arm/Group | Arm A (Palonosetron 0.25 mg IV on Day 1) | Arm B (Ondansetron 24 mg Oral on Day 1)
Started | 20 | 20
Overall Complete Response Rate | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Palonosetron 0.25 mg day 1; aprepitant 125 mg day 1, 80 mg day 2-3; dexamethasone 12 mg day 1, 8 mg day 2-4
- Arm B: Ondansetron 24 mg day 1; aprepitant 125 mg day 1, 80 mg day 2-3; dexamethasone 12 mg day 1, 8 mg day 2-4
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 32
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Overall CR(Complete Response)After the First Course of HEC, Defined as no Emesis and no Use of Rescue Medication
Description: We will use exact binomial methods to estimate proportions and their associated 95% confidence intervals.
Time Frame: Up to 120 hours after completion of chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Arm A (Palonosetron 0.25 mg IV on Day 1): Palonosetron 0.25 mg IV once on day 1, 30 minutes prior to chemotherapy, aprepitant 125 mg orally once on day 1, 60 minutes prior to chemotherapy, then 80 mg once daily on days 2 and 3 at the same time, and dexamethasone 12 mg orally once on day 1, 30 minutes prior to chemotherapy, then 8 mg once daily on days 2 through 4.
- Arm B (Ondansetron 24 mg Oral on Day 1): Ondansetron 24 mg once orally on day 1, 30 minutes prior to chemotherapy, aprepitant 125 mg orally once on day 1, 60 minutes prior to chemotherapy, then 80 mg once daily on days 2 and 3, and dexamethasone 12 mg orally once on day 1, 30 minutes prior to chemotherapy, then 8 mg once daily on days 2 through 4.
Arm/Group | Arm A (Palonosetron 0.25 mg IV on Day 1) | Arm B (Ondansetron 24 mg Oral on Day 1)
Number analyzed (Participants) | 20 | 20
percentage of patients | 65 [40.8 to 84.6] | 40 [19.1 to 63.9]

2. Secondary Outcome: Acute CR (Complete Response)
Description: After the First Course of HEC, Defined as no Emesis and no Use of Rescue Medication from time 0 to 24 hours.
Time Frame: 0-24 hours after chemotherapy
Measure: Number; unit: percentage of particpants
Arm/Group | Arm A (Palonosetron 0.25 mg IV on Day 1) | Arm B (Ondansetron 24 mg Oral on Day 1)
Number analyzed (Participants) | 20 | 20
percentage of particpants | 75 | 55

3. Secondary Outcome: Delayed CR (Complete Response)
Description: After the First Course of HEC, Defined as no Emesis and no Use of Rescue Medication From Time 24to 120 Hours.
Time Frame: 24-120 hours after chemotherapy
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Palonosetron 0.25 mg IV on Day 1) | Arm B (Ondansetron 24 mg Oral on Day 1)
Number analyzed (Participants) | 20 | 20
percentage of participants | 65 | 45

4. Secondary Outcome: Percentage of Patients Who Experienced Grade 1, 2 or 3 Nausea From Time 0 to 120 Hours
Description: The percentage of patients who experienced grade 1, 2 or 3 nausea from time 0 to 120 hours. Nausea graded using the National Cancer Institute (NCI) CTCAE (Common Toxicity Criteria for Adverse Effects)version 4.0 Nausea Grading Scale. Grade 1=Loss of appetite without alteration in eating habits, Grade 2= Oral intake decreased without significant weight loss, dehydration or malnutrition, Grade 3= Inadequate oral caloric or fluid intake; tube feeding, TPN, or hospitalization indicated.
Time Frame: Time 0 to 120 hours
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Palonosetron 0.25 mg IV on Day 1) | Arm B (Ondansetron 24 mg Oral on Day 1)
Number analyzed (Participants) | 20 | 20
percentage of participants | 55 | 65

5. Secondary Outcome: Visual Analog Scale (VAS) Scores
Time Frame: Up to 7 days after completion of study treatment
Population: VAS Scores were not collected
Arm/Group | Arm A (Palonosetron 0.25 mg IV on Day 1) | Arm B (Ondansetron 24 mg Oral on Day 1)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Use of Rescue Medication for Each Treatment Arm
Time Frame: From time 0 to 120 hours
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Palonosetron 0.25 mg IV on Day 1) | Arm B (Ondansetron 24 mg Oral on Day 1)
Number analyzed (Participants) | 20 | 20
percentage of participants | 35 | 55

7. Secondary Outcome: Percentage of Patients Who Experienced Grade 1, 2 or 3 Vomiting From Time 0 to 120 Hours
Description: The percentage of patients who experienced grade 1, 2 or 3 vomiting from time 0 to 120 hours. Nausea graded using the National Cancer Institute (NCI) CTCAE v 4.0 vomiting Grading Scale. Grade 1=Loss of appetite without alteration in eating habits, Grade 2= Oral intake decreased without significant weight loss, dehydration or malnutrition, Grade 3= Inadequate oral caloric or fluid intake; tube feeding, TPN, or hospitalization indicated.
Time Frame: From time 0 to 120 hours
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Palonosetron 0.25 mg IV on Day 1) | Arm B (Ondansetron 24 mg Oral on Day 1)
Number analyzed (Participants) | 20 | 20
percentage of participants | 5 | 15

ADVERSE EVENTS:
Time Frame: Days 1 through 5 following chemotherapy
Description: Patients were given a diary on the day of treatment to record symptoms experienced on days 1 through 6. Although symptoms were documented on days 1 through 6, they were only evaluated based upon days 1 through 5. The additional day of recording was instituted to ensure the investigators captured the entire day 1 through time period.
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=20) | Arm B (N=20)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No